CLINICAL TRIAL: NCT02070874
Title: Palliative Care Symptom Management in Rural Communities
Brief Title: Pain and Symptom Management in Rural Communities
Acronym: TelePain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Ardith Doorenbos, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00002019; R01NR012450 (NIH)
Record Dates: First submitted 2014-02-20; First posted 2014-02-25 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Chronic Pain; Palliative Care
Keywords: pain and symptom management
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- telehealth enhanced pain management (Experimental): video-case conferences for providers PainTracker for patients
  Interventions: Behavioral: telehealth enhanced pain management
- usual care (No Intervention): usual care

INTERVENTIONS:
Behavioral: telehealth enhanced pain management
  Arms: telehealth enhanced pain management

SUMMARY:
Patients in isolated rural settings often lack easy access to pain care and specialist services. Yet rural residents are more likely than their urban counterparts to be older; be in poorer overall health; suffer from more chronic or serious illnesses and disabilities; be uninsured or underinsured; and live in poverty. Telehealth is an emerging method of health care delivery that has been found useful and effective in many clinical settings and specialties. Telehealth technologies can bridge geographic distance and increase access to specialist care in rural settings. The investigators propose a cluster randomized clinical trial design to test the effects of a telehealth-enhanced palliative care pain-management program for 240 patients and 40 providers in rural health care settings. The proposed program will provide services to both patients and providers: Patients will conduct self-assessments and report pain and other symptoms via telehealth. Health care providers will receive telehealth-delivered case consultations that will include case management, evidence-based practice resources, and peer support. Providers and their patients will be randomly assigned to intervention groups, which receive the telehealth-enhanced palliative care pain-management intervention, or to control groups. The investigators primary aim is to compare patient self-reports of pain and quality of life in the intervention and control groups over 2 months. Aim 2 is to examine, in the intervention and control groups over 2 months, providers' knowledge and attitudes regarding pain and perceived competence in treating pain. Aim 3 is to evaluate the cost-effectiveness of the telehealth intervention. The investigators will use mixed effects models with patients nested within providers to evaluate the effect of the intervention on study outcomes. Findings from this study will be instrumental in advancing telehealth and improving pain management and palliative care among underserved rural populations.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* diagnosed with pain
* completion of an outpatient visit in the past 2 months
* functional fluency in English
* no cognitive impairment
* no problems with regular phone lines

Exclusion Criteria:

-

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
pain | 12 weeks
  pain severity

SECONDARY OUTCOMES:
PHQ 4 | 12 weeks
  anxiety and depressive symptoms

OTHER OUTCOMES:
cost | 12 weeks
  HUI-3

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bensink ME, Eaton LH, Morrison ML, Cook WA, Curtis RR, Gordon DB, Kundu A, Doorenbos AZ. Cost effectiveness analysis for nursing research. Nurs Res. 2013 Jul-Aug;62(4):279-85. doi: 10.1097/NNR.0b013e318298b0be. PMID 23817285
- [Background] Eaton LH, Gordon DB, Wyant S, Theodore BR, Meins AR, Rue T, Towle C, Tauben D, Doorenbos AZ. Development and implementation of a telehealth-enhanced intervention for pain and symptom management. Contemp Clin Trials. 2014 Jul;38(2):213-20. doi: 10.1016/j.cct.2014.05.005. Epub 2014 May 17. PMID 24846620
- [Result] Theodore BR, Whittington J, Towle C, Tauben DJ, Endicott-Popovsky B, Cahana A, Doorenbos AZ. Transaction cost analysis of in-clinic versus telehealth consultations for chronic pain: preliminary evidence for rapid and affordable access to interdisciplinary collaborative consultation. Pain Med. 2015 Jun;16(6):1045-56. doi: 10.1111/pme.12688. Epub 2015 Jan 23. PMID 25616057
- [Result] Meins AR, Doorenbos AZ, Eaton L, Gordon D, Theodore B, Tauben D. TelePain: A Community of Practice for Pain Management. J Pain Relief. 2015 Mar 11;4(2):177. doi: 10.4172/2167-0846.1000177. PMID 25964869